CLINICAL TRIAL: NCT02438332
Title: Retrospective Study of Reoperation After Primary Augmentation With NATRELLE® INSPIRA® Breast Implants
Acronym: RANBI-I
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-CAN-PLS-0337
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Breast Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- NATRELLE® INSPIRA® TruForm® 1 (Smooth): Subjects receiving primary breast augmentation with smooth NATRELLE® INSPIRA® TruForm® 1 breast implants
  Interventions: Device: Smooth NATRELLE® INSPIRA® TruForrm® 1 Breast Implants
- NATRELLE® INSPIRA® TruForm® 1 (Textured): Subjects receiving primary breast augmentation with textured NATRELLE® INSPIRA® TruForm® 1 breast implants
  Interventions: Device: Textured NATRELLE® INSPIRA® TruForm® 1 Breast Implants
- NATRELLE® INSPIRA® TruForm® 2 (Smooth): Subjects receiving primary breast augmentation with smooth NATRELLE® INSPIRA® TruForm® 2 breast implants
  Interventions: Device: Smooth NATRELLE® INSPIRA® TruForrm® 2 Breast Implants
- NATRELLE® INSPIRA® TruForm® 2 (Textured): Subjects receiving primary breast augmentation with textured NATRELLE® INSPIRA® TruForm® 2 breast implants
  Interventions: Device: Textured NATRELLE® INSPIRA® TruForm® 1 Breast Implants

INTERVENTIONS:
Device: Smooth NATRELLE® INSPIRA® TruForrm® 1 Breast Implants — Surgical implant
  Other Names: Round cohesive, gel-filled breast implants (low, low plus, moderate, full, or extra full projection)
  Groups: NATRELLE® INSPIRA® TruForm® 1 (Smooth)
Device: Textured NATRELLE® INSPIRA® TruForm® 1 Breast Implants — surgical implant
  Other Names: Round cohesive, gel-filled breast implants (low, low plus, moderate, full, or extra full projection)
  Groups: NATRELLE® INSPIRA® TruForm® 1 (Textured)
Device: Smooth NATRELLE® INSPIRA® TruForrm® 2 Breast Implants — surgical implant
  Other Names: Round cohesive, gel-filled breast implants (low, low plus, moderate, full, or extra full projection)
  Groups: NATRELLE® INSPIRA® TruForm® 2 (Smooth)
Device: Textured NATRELLE® INSPIRA® TruForm® 1 Breast Implants — surgical implant
  Other Names: Round cohesive, gel-filled breast implants (low, low plus, moderate, full, or extra full projection)
  Groups: NATRELLE® INSPIRA® TruForm® 2 (Textured)

SUMMARY:
This study will evaluate the incidence of reoperations associated with the use of smooth and textured NATRELLE® INSPIRA® TruForm® 1 and TruForm® 2 devices in patients who have undergone primary breast augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Primary breast augmentation (either bilateral or unilateral) operated on by the investigating surgeon with an infra-mammary approach smooth or textured NATRELLE® INSPIRA® TruForm® 1 or 2 device
* Primary breast augmentation 2 to 4 years (24-48 months) prior to data collection
* Subfascial, submuscular, dual plane or subglandular implant placement

Exclusion Criteria:

* Breast augmentation for Poland Syndrome or amastia
* Breast reconstruction following mastectomy
* Revision or secondary breast reconstruction
* Non NATRELLE® INSPIRA® device implanted at initial breast augmentation
* Women diagnosed with breast disease considered to be pre-malignant or malignant prior to or at the time of primary breast augmentation
* Surgical procedures of the breast not related to the primary breast augmentation (e.g. excision of significant skin lesions or a biopsy) occurring prior to or at the time of primary augmentation that may adversely affect the aesthetic outcome in the opinion of the investigator
* Axillary or peri-areolar approach
* Mastopexy augmentation

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that have undergone a primary breast augmentation for aesthetic reasons with NATRELLE® INSPIRA® TruForm® 1 or TruForm® 2 implant.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2014-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Reoperations of All Cause Following the Use of Smooth or Textured NATRELLE® INSPIRA® TruForm® 1 or TruForm® 2 Breast Implants | 4 Years

SECONDARY OUTCOMES:
Incidence (by Product Type) of First Reoperation Following the Use of Smooth or Textured NATRELLE® INSPIRA® TruForm®1 or TruForm® 2 Breast Implants | 4 Years
Reasons For Primary Augmentation | 4 Years
Time From the Date of Implant Until First Reoperation | 4 Years
Reasons For Reoperation Incidence | 4 Years
Incidences of Implant Removal With Replacement | 4 Years
Incidences of Implant Removal Without Replacement | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (17):
- Canada (17):
  - Banff Plastic Surgery, Banff, Alberta
  - Macleod Trail Plastic Surgery, Calgary, Alberta
  - Jonathan Toy, Edmonton, Alberta
  - Y.E.S MedSpa & Cosmetic Surgery Centre, Langley, British Columbia
  - Institute of Cosmetic and Laser Surgery, Oakville, Ontario
  - Ottawa Plastic Surgery: Dr. Howard Silverman, Ottawa, Ontario
  - Rice Cosmetic Surgery, Toronto, Ontario
  - Cosmedical Rejuvenation Clinic, Toronto, Ontario
  - Yorkville Institute of Plastic Surgery, Toronto, Ontario
  - SpaSurgica, Waterloo, Ontario
  - Centre de Medecine et de Chirurgie Ambulatoires Isomed, Boucherville, Quebec
  - CCPEM, Montreal, Quebec
  - Cosmedica, Pointe-Claire, Quebec
  - Clinique de Chirurgie Plastique et Esthétique de la Haute-Ville, Québec, Quebec
  - Sebastien Nguyen MD Inc., Québec, Quebec
  - Cosmetic Surgery Clinic, Waterloo, Quebec
  - Sandra McGill MD Inc., Westmount, Quebec